CLINICAL TRIAL: NCT03841084
Title: Blend to Limit oxygEN in ECMO: a ranDomised controllEd Registry Trial The BLENDER Trial - A Phase II Multicentre Randomised Controlled Trial
Brief Title: Blend to Limit Oxygen in ECMO: A Randomised Controlled Registry Trial
Acronym: BLENDER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZIC-RC/DP001
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Failure; Critical Illness
Keywords: ECMO; V-A ECMO; Oxygen; Hyperoxia
MeSH Terms: conditions — Heart Failure; Critical Illness; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: This is a phase II, registry-based, multicentre, parallel group randomised controlled trial.
  (Data retrieved from the EXCEL national clinical registry)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conservative Oxygen Management Strategy (Active Comparator): Patients allocated to the conservative strategy will have the ECMO blender oxygen fraction (FbO2) will be titrated to achieve a post-oxygenator saturations of 92-96% (the FbO2 cannot be reduced to lower than 0.5). Post-oxygenator arterial blood gases (ABG's) will be taken to ensure safety and to allow for adjustments to be made. The ventilator FiO2 will be titrated to patient oxygen saturations (SpO2) of 92-96%.
  Interventions: Drug: Oxygen
- Liberal Oxygen Management Strategy (Active Comparator): Patients allocated to the liberal strategy will have the FbO2 set at 1.0 at all times. The ventilator FiO2 will be titrated to achieve a patient oxygen saturations (SpO2) of 97-100% (but not lower than 0.5).
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Conservative oxygen management strategy- reduces oxygen on the inoblender in the ECMO circuit.
  Liberal oxygen management strategy - does not reduce the oxygen on the inoblender via the ECMO circuit

SUMMARY:
To determine in patients requiring venoarterial (V-A) ECMO, whether the use of a conservative as compared with liberal oxygen strategy, results in a greater number of ICU-free days at day 28.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) can be a lifesaving procedure for the sickest patients in the Intensive Care Unit (ICU) who are at risk of death from severe cardiac and respiratory failure. ECMO is a device which pumps blood out of the body and returns it back after adding oxygen and removing carbon dioxide. While potentially life-saving, ECMO is associated with high use of critical care resources and increased risk of adverse outcomes in survivors.

The BLENDER Trial is a multicentre trial in ECMO patients to determine whether a conservative oxygen strategy during ECMO reduces ICU length of stay and improves patient outcomes compared to a liberal oxygen strategy. Both strategies are currently standard practice worldwide, however, there is no consensus to which strategy is better for our patients. This trial aims to utilise an existing intensive care registry and will recruit 300 patients with life threatening acute cardiac or respiratory failure. If the BLENDER Trial confirms that one oxygen management strategy is more effective than the other, its findings may improve the lives of critically ill Australians and inform clinical practice worldwide.

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥18 years who are commenced on V-A ECMO for severe cardiac, or following refractory cardiac arrest.

Exclusion Criteria:

* Greater than 6 hours have elapsed from the time of initiation of ECMO to randomisation
* Patients who are suspected or confirmed to be pregnant
* Where an indication exists for a specific oxygen target as part of clinical care (e.g. carbon monoxide poisoning)
* Patients who are already enrolled in another oxygen titration study (unless agreed by study committees)
* Patients not willing to receive blood products (e.g. Jehovah's Witness)
* Where the treating physician deems the study is not in the patient's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the number of alive and ICU-free days to day 28. | at day 28
  ICU free days are defined as the total number of days (or part days) being free of ICU between randomisation and day 28, with the exception that all patients who die by day 28 will be defined as having zero ICU free days.

SECONDARY OUTCOMES:
Hospital mortality | at day 28
  Mortality rates of patients that day in hospital from randomisation to day 28
ICU mortality | at day 28
  Mortality rates of patients that day in ICU from randomisation to day 28
ICU length of stay | at day 28
  Number of hours spent in ICU from randomisation up to day 28
Duration of mechanical ventilation | at day 28
  Number of hours requiring mechanical ventilation from randomisation to day 28
Disability | 6 and 12 months
  World Health Organisation's Disability Assessment Schedule 2.0 12L
Health-related quality of life at six and twelve months using the EQ5D-5L | 6 and 12 months
  Euro Qol Group Health Survey (EQ-5D-5L) Measuring quality of life which looks at five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Psychological function at six and twelve months | 6 months & 12 months
  Measured using a trained, blinded assessor via telephone interview

OTHER OUTCOMES:
ECMO circuit life | day 28
  number of hours that each circuit was in use

CONTACTS AND LOCATIONS:
Overall Officials: David Pilcher, Principal Investigator — Monash University, Australian & New Zealand Intensive Care research Centre
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gu WJ, Shi R, Cen Y, Ye YY, Xie XD, Yin HY. Association Between Arterial Hyperoxia and Mortality in Pediatric and Adult Patients Undergoing Extracorporeal Membrane Oxygenation: A Systematic Review and Meta-Analysis. Anesth Analg. 2025 Jun 1;140(6):1367-1376. doi: 10.1213/ANE.0000000000007348. Epub 2024 Dec 20. PMID 39705180
- [Derived] Burrell A, Ng S, Ottosen K, Bailey M, Buscher H, Fraser J, Udy A, Gattas D, Totaro R, Bellomo R, Forrest P, Martin E, Reid L, Ziegenfuss M, Eastwood G, Higgins A, Hodgson C, Litton E, Nair P, Orford N, Pellegrino V, Shekar K, Trapani T, Pilcher D. Blend to Limit OxygEN in ECMO: A RanDomised ControllEd Registry (BLENDER) Trial: Study Protocol and Statistical Analysis Plan. Crit Care Resusc. 2023 Aug 4;25(3):118-125. doi: 10.1016/j.ccrj.2023.06.001. eCollection 2023 Sep. PMID 37876374
- [Derived] Joyce CJ, Anderson C, Shekar K. Hyperoxia on Venoarterial Extracorporeal Membrane Oxygenation: A Modifiable Risk? Crit Care Med. 2022 Jan 1;50(1):e99-e100. doi: 10.1097/CCM.0000000000005252. No abstract available. PMID 34914658